CLINICAL TRIAL: NCT00566319
Title: A Randomised Controlled Trial to Investigate the Effect of a Structured Educational Programme on Physical Activity Levels and Glucose Tolerance in People With Impaired Glucose Tolerance
Brief Title: Can Structured Education Promote Physical Activity in Those Identified With an Increased Risk of Developing Diabetes
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Prof. Melanie Davies, University of Leicester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 06/Q2502/29; BDA:RD05/0003159
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Prediabetic State
Keywords: Exercise
MeSH Terms: conditions — Prediabetic State; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: PREPARE with pedometer
- 2 (Active Comparator)
  Interventions: Behavioral: PREPARE

INTERVENTIONS:
Behavioral: PREPARE with pedometer — Structured educational programme with pedometer use
  Arms: 1
Behavioral: PREPARE — Structured educational programme
  Arms: 2

SUMMARY:
This study is a three-armed randomised controlled trial that aims to determine the effect of a structured educational programme on physical activity levels and glucose tolerance in individuals with impaired glucose tolerance (IGT). The educational programme is designed to promote physical activity by targeting perceptions and knowledge of IGT, exercise self-efficacy, and self-regulatory skills. The study will also investigate whether the effectiveness of the educational programme at promoting self-regulatory skills and physical activity is enhanced by the inclusion of a pedometer and personalised step/day goals.

ELIGIBILITY:
Inclusion Criteria:

* 2-h blood glucose ≥ 7.8 mmol/l and < 11.1 mmol/l
* Fasting plasma glucose < 7 mmol/l
* BMI ≥ 25 kg/m2 (or 23 kg/m2 for those from a South Asian ethnic origin)
* Aged 18 or over

Exclusion Criteria:

* Taking medication known to significantly interfere with glucose tolerance
* Participating in regular vigorous physical activity
* Unable to participate in moderate intensity physical activity
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-10; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
2-hour glucose | 2 hours

SECONDARY OUTCOMES:
Pedometer counts, Fasting glucose, total cholesterol, HDL-cholesterol, LDL- cholesterol, TNFα, IL-6, CRP, systolic and diastolic blood pressure, body mass, waist circumference, BMI, physical activity, psychological determinants | Pedometer counts, 7 days ; everything else, 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Davies, MD, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, Leicester, United Kingdom

REFERENCES:
- [Derived] Yates T, Davies MJ, Sehmi S, Gorely T, Khunti K. The Pre-diabetes Risk Education and Physical Activity Recommendation and Encouragement (PREPARE) programme study: are improvements in glucose regulation sustained at 2 years? Diabet Med. 2011 Oct;28(10):1268-71. doi: 10.1111/j.1464-5491.2011.03357.x. PMID 21672008